CLINICAL TRIAL: NCT00863590
Title: A Double-Blind, Randomized, Placebo-Controlled, Multi-Panel, Single Oral Rising-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of MK0822 in Healthy Volunteers
Brief Title: A Single-Dose Study of the Safety, Tolerability, and Pharmacokinetics of Odanacatib (MK0822) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-001; 2009_562
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- A (Experimental): Panel A
  Interventions: Drug: odanacatib
- B (Experimental): Panel B
  Interventions: Drug: Comparator: odanacatib (Panel B)
- C (Experimental): Panel C
  Interventions: Drug: Comparator: odanacatib (Panel C)
- D (Experimental): Panel D
  Interventions: Drug: Comparator: odanacatib (Panel D)

INTERVENTIONS:
Drug: odanacatib — [Intervention Name: odanacatib (Panel A)] Panel A: Odanacatib tablets will be administered to male subjects in rising single doses of 2, 10, 50, 200, or 400 mg over 5 treatment periods. Each subject will receive placebo to odanacatib in one or two of the 5 treatment periods. There will be at least 7 days between each treatment period.
  Arms: A
Drug: Comparator: odanacatib (Panel B) — Panel B: Odanacatib tablets will be administered to male subjects in rising single doses of 5, 25 (fasting), 100, 25 (fed), or 600 mg over 5 treatment periods. Each subject will receive placebo to odanacatib in one or two of the 5 treatment periods. There will be at least 7 days between each treatment period.
  Arms: B
Drug: Comparator: odanacatib (Panel C) — Panel C: Odanacatib tablets will be administered to female subjects in rising single doses of 50 or 100 mg over 2 treatment periods. Half of the subjects will receive placebo to odanacatib in one of the 2 treatment periods. There will be at least 7 days between each treatment period.
  Arms: C
Drug: Comparator: odanacatib (Panel D) — Panel D: Odanacatib tablets or placebo to odancatib will be administered to male subjects in rising single doses of 100, 200, or 300 mg following a high-fat breakfast over 3 treatment periods. Three of twelve subjects will receive placebo to odanacatib in all 3 treatment periods. There will be at least 10 days between each treatment period.
  Arms: D

SUMMARY:
This study assessed the safety, tolerability, and pharmacokinetics of single-dose odanacatib (MK0822) with and without food.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is a male between the ages of 18 and 45 years or (for Part I only) a female 60 years or younger
* Female subject is postmenopausal
* Subject is within 20% of ideal body weight
* Subject is a nonsmoker

Exclusion Criteria:

* Subject has multiple or severe allergies to food or medications
* Subject has a history of metabolic bone disease, kidney/bladder stones, or treatment with bisphosphonates
* Subject has any infections, including HIV
* Subject consumes excessive amounts of caffeine or alcohol
* Subject has donated blood or taken another investigational drug in the last month
* Subject has a history of any illness that may confound the results of the study or pose additional risk in administering the study drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-06; Primary Completion 2005-02 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
safety and tolerability based on assessment of clinical and laboratory adverse experiences | Part I: 12 Weeks, Part II: 13 Weeks

SECONDARY OUTCOMES:
Plasma concentration of MK0822 | Up to 336 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Stoch SA, Zajic S, Stone JA, Miller DL, van Bortel L, Lasseter KC, Pramanik B, Cilissen C, Liu Q, Liu L, Scott BB, Panebianco D, Ding Y, Gottesdiener K, Wagner JA. Odanacatib, a selective cathepsin K inhibitor to treat osteoporosis: safety, tolerability, pharmacokinetics and pharmacodynamics--results from single oral dose studies in healthy volunteers. Br J Clin Pharmacol. 2013 May;75(5):1240-54. doi: 10.1111/j.1365-2125.2012.04471.x. PMID 23013236